CLINICAL TRIAL: NCT00007501
Title: CSP #403 - Trial of Varicella Zoster Vaccine for the Prevention of Herpes Zoster and Its Complications
Brief Title: Shingles Prevention Study
Acronym: SPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 403; NCT00001907 (obsolete NCT alias); NCT00006065 (obsolete NCT alias); NCT00006069 (obsolete NCT alias); NCT00023257 (obsolete NCT alias)
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Herpes Zoster; Postherpetic Neuralgia
Keywords: varicella-zoster vaccine
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): varicella-zoster vaccine
  Interventions: Biological: Varicella-zoster vaccine
- Arm 2 (Placebo Comparator): vaccine placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Varicella-zoster vaccine — Immunization with 0.5 ml, live, attenuated (Oka/Merck) varicella-zoster vaccine.
  Arms: Arm 1
Biological: Placebo — Placebo vaccine
  Arms: Arm 2

SUMMARY:
The incidence and severity of HZ (or shingles), as well as the frequency and severity of its complications, increases markedly with increasing age. More than half of all cases occur in persons over the age of 60. Even without complications, HZ can interfere with an elderly patient's ability to perform essential activities of daily living, resulting in a loss of independence that is emotionally devastating and frequently irreversible. The most common complication of HZ in elderly persons is postherpetic neuralgia (PHN), which frequently results in disordered sleep, chronic fatigue, anxiety and severe depression. Antiviral therapy has a modest impact on the acute phase of HZ. However, it does not appear to prevent the development of PHN.

This study is a 5.5 year randomized, double-blind, placebo-controlled, efficacy trial to determine whether vaccination with live-attenuated Oka/Merck varicella-zoster decreases the incidence and/or severity of herpes zoster (HZ) and its complications in adults 60 years of age and older.

DETAILED DESCRIPTION:
Primary Hypothesis:

Immunization with live, attenuated (Oka/Merck) varicella-zoster vaccine will significantly reduce the burden of illness associated with herpes zoster (HZ).

Secondary Hypotheses:

Immunization with live, attenuated (Oka/Merck) varicella-zoster vaccine will reduce the incidence of postherpetic neuralgia (PHN).

Primary Outcomes:

The primary outcome is the burden of illness due to HZ defined by the area under the worst pain versus time curve measured during the 6 month period following HZ rash onset in subjects who develop of HZ. The burden of illness outcome is sensitive to the incidence, severity, and duration of HZ-associated pain. The secondary outcome is the incidence of PHN, where PHN is defined as HZ-associated pain rated as greater than or equal to 3 (on a 0 to 10 scale) persisting or appearing more than 30 days after the onset of the HZ rash.

Interventions:

Immunization with 0.5 ml, live, attenuated (Oka/Merck) varicella-zoster vaccine versus vaccine placebo.

Study Abstract:

The incidence and severity of HZ (or shingles), as well as the frequency and severity of its complications, increases markedly with increasing age. More than half of all cases occur in persons over the age of 60. Even without complications, HZ can interfere with an elderly patient's ability to perform essential activities of daily living, resulting in a loss of independence that is emotionally devastating and frequently irreversible. The most common complication of HZ in elderly persons is postherpetic neuralgia (PHN), which frequently results in disordered sleep, chronic fatigue, anxiety and severe depression. Antiviral therapy has a modest impact on the acute phase of HZ. However, it does not appear to prevent the development of PHN.

This study was a 5.5 year randomized, double-blind, placebo-controlled, efficacy trial to determine whether vaccination with live-attenuated Oka/Merck varicella-zoster decreases the incidence and/or severity of herpes zoster (HZ) and its complications in adults 60 years of age and older; 37,200 subjects over 60 years of age will be randomized at 22 sites to receive either vaccine or placebo. At least one third of the subjects were to be 70 years of age or older. Subjects were followed actively for HZ until at least 750 cases of HZ and at least 62 cases of PHN occurred. Subjects who developed HZ were evaluated for severity and duration of associated pain, extent and duration of rash, and for changes in quality of life associated with the disease for six months after the onset of HZ rash. All adverse events (serious and non-serious) occurring within 42 days after vaccination were recorded. Thereafter, serious adverse events were recorded if assessed as possibly related to the vaccination. An adverse event substudy was to enroll 6000 subjects for recording all adverse events on a vaccination Report Card. Substudy participants were also followed for any hospital admissions during the study.

The study was initiated in December 1998. Patient recruitment began in November 1998 at one site, at 20 sites between February 1999 and July 1999, and at one site that was added in January 2000. On September 26, 2001, enrollment in the study was completed with 38,456 randomized subjects. The time point for the study definition of PHN was changed by protocol amendment from 30 days to 90 days after HZ rash onset. A formal sample size re-estimation was performed in June 2003. The Executive Committee and DSMB reviewed these results and approved the increase in event size from 400 to 750 evaluable cases of HZ for the primary endpoint. It was projected that the number of evaluable cases of HZ for the primary endpoint and the number of evaluable cases of PHN for the secondary (co-primary) endpoint would be observed by the end of September 2003. Therefore, the Study initiated its closeout plan beginning in October 2004. Follow-up of the last suspected case of HZ was completed in March 2004 and closeout interviews for the more than 37,000 surviving subjects were completed as of April 28, 2004.

The results of the main efficacy and safety analyses were unblinded on December 1, 2004, and presented to the DSMB, Executive Committee, and representatives for Merck & Co., Inc. Letters were sent to the study subjects informing them of the overall results and the treatment they received. The main manuscript was published in the New England Journal of Medicine (June 2005; 352:2271-84). The vaccine was approved for the prevention of shingles by the FDA on May 25, 2006. The main efficacy study is closed. Additionally, three substudies have been conducted:

A substudy (CSP#403B) was initiated in November 2005 to offer investigational zoster vaccine to the placebo recipients of CSP#403. Vaccination was completed in March 2007 with 13,681 (75%) of the placebo recipients vaccinated. This substudy is closed. The safety results from the substudy were published in the Journal of Infectious Diseases (J Infect Dis. 2013 May 31 epub).

A short-term persistence substudy (CSP#403A) was initiated in September 2004 to extend the follow-up vaccine and placebo recipients to assess the longer term effectiveness of the vaccine. This substudy bridged the period between the end of the efficacy study and the vaccination of placebo recipients and the initiation of a long-term persistence study. The study enrolled 14,270 subjects and completed follow-up in May 2007. This substudy is closed and is in ongoing analysis. The primary results for this study were published in Clinical Infectious Diseases (Clin Infect Dis. 2012 Nov 15;55(10):1320-1328)

CSP#403C, the Long-Term Persistence Substudy, was initiated in March 2006 and enrolled 6867 vaccine recipients from the main efficacy study. Enrollment was restricted to vaccine recipients from the main efficacy study with no history of herpes zoster. This study was initiated to complete an additional five-years of follow-up post-vaccination. The objective of this study was to estimate the longer-term durability of zoster vaccine efficacy by following a cohort of vaccine recipients from the primary efficacy study for three study outcomes: 1) the incidence of herpes zoster, 2) the incidence of postherpetic neuralgia (PHN), and 3) the burden of illness (BOI) due to herpes zoster. The study completed surveillance for new cases of herpes zoster as of December 2010 and completed the follow-up of the last case of herpes zoster in February 2011. All study sites have been closed out. This substudy has been completed and is in the final analysis phase.

ELIGIBILITY:
Inclusion Criteria:

* Adults 60 years of age and older.
* History of Chickenpox.
* Have given written informed consent prior to enrollment.
* History of varicella or long-term (greater than or equal to 30 years) residence in the continental USA.

Exclusion Criteria:

* No history of shingles, no current history of immune suppression (e.g. malignancy or neoplastic disease, corticosteroid therapy).
* No immunosuppression resulting from disease (e.g., malignancy; HIV infection), corticosteroids (except intermittent topical or inhaled corticosteroid [greater than 800 mcg/day beclomethasone dipropionate or equivalent]), or other immunosuppressive/cytotoxic therapy (cancer chemotherapy or organ transplantation).
* No active neoplastic disease (except local skin cancer or other malignancies [e.g., prostate cancer] that are stable in the absence of immunosuppressive/cytotoxic therapy).
* No prior Herpes Zoster.
* No prior receipt of varicella vaccine.
* No allergic sensitivity to neomycin.
* No history of anaphylactoid reaction to gelatin.
* No significant underlying illness that would be expected to prevent completion of the study (e.g., life-threatening disease likely to limit survival to less than 5 years).
* Not ambulatory (must not be bed-ridden or homebound).
* No receipt of immune globulin or any other blood product within 3 months before or planned during the 3-5 year study period.
* No receipt of any other immunizations within one month before study vaccination (2 weeks in the case of inactivated influenza vaccines or other non-replicating immunization products [e.g., dT, pneumococcal vaccine, hepatitis A vaccine, hepatitis B vaccine]), or scheduled within 6 weeks after study vaccination.
* Not currently receiving antiviral therapy.
* No other condition (e.g., extensive psoriasis, chronic pain syndrome, cognitive impairment, severe hearing loss) that, in the opinion of the investigator, might interfere with the evaluations required by the study.
* No intercurrent illness (e.g., urinary tract infection, influenza) that might interfere with the interpretation of the study.
* No females who are pre-menopausal.
* No subjects unlikely to adhere to protocol follow-up.
* No subjects involved in a conflicting (vaccine or investigational drug) clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38456 (Actual)
Dates: Start 1998-11; Primary Completion 2004-04 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Reduce burden of illness due to herpes zoster (HZ) | Incidence of postherpetic neuralgia (PHN), where PHN is defined as HZ-associated pain greater than or equal to 3 persisting or appearing more than 30 days after the onset of the HZ rash

CONTACTS AND LOCATIONS:
Overall Officials: Michael N. Oxman, Study Chair — VA San Diego Healthcare System, San Diego
Locations (22):
- United States (22):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - University of Colorado, Denver, Colorado
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Medical Center, Lexington, Lexington, Kentucky
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - NIH-NIAID (Bethesda, MD), Bethesda, Maryland
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, St Louis, St Louis, Missouri
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Northport, Northport, New York
  - Rochester, NY (NIH), Rochester, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor University, Houston, Texas
  - University of Texas at San Antonio, San Antonio, Texas
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

REFERENCES:
- [Result] Oxman MN, Levin MJ, Johnson GR, Schmader KE, Straus SE, Gelb LD, Arbeit RD, Simberkoff MS, Gershon AA, Davis LE, Weinberg A, Boardman KD, Williams HM, Zhang JH, Peduzzi PN, Beisel CE, Morrison VA, Guatelli JC, Brooks PA, Kauffman CA, Pachucki CT, Neuzil KM, Betts RF, Wright PF, Griffin MR, Brunell P, Soto NE, Marques AR, Keay SK, Goodman RP, Cotton DJ, Gnann JW Jr, Loutit J, Holodniy M, Keitel WA, Crawford GE, Yeh SS, Lobo Z, Toney JF, Greenberg RN, Keller PM, Harbecke R, Hayward AR, Irwin MR, Kyriakides TC, Chan CY, Chan IS, Wang WW, Annunziato PW, Silber JL; Shingles Prevention Study Group. A vaccine to prevent herpes zoster and postherpetic neuralgia in older adults. N Engl J Med. 2005 Jun 2;352(22):2271-84. doi: 10.1056/NEJMoa051016. PMID 15930418
- [Result] Simberkoff MS, Arbeit RD, Johnson GR, Oxman MN, Boardman KD, Williams HM, Levin MJ, Schmader KE, Gelb LD, Keay S, Neuzil K, Greenberg RN, Griffin MR, Davis LE, Morrison VA, Annunziato PW; Shingles Prevention Study Group. Safety of herpes zoster vaccine in the shingles prevention study: a randomized trial. Ann Intern Med. 2010 May 4;152(9):545-54. doi: 10.7326/0003-4819-152-9-201005040-00004. PMID 20439572
- [Result] Levin MJ, Oxman MN, Zhang JH, Johnson GR, Stanley H, Hayward AR, Caulfield MJ, Irwin MR, Smith JG, Clair J, Chan IS, Williams H, Harbecke R, Marchese R, Straus SE, Gershon A, Weinberg A; Veterans Affairs Cooperative Studies Program Shingles Prevention Study Investigators. Varicella-zoster virus-specific immune responses in elderly recipients of a herpes zoster vaccine. J Infect Dis. 2008 Mar 15;197(6):825-35. doi: 10.1086/528696. PMID 18419349
- [Result] Harbecke R, Oxman MN, Arnold BA, Ip C, Johnson GR, Levin MJ, Gelb LD, Schmader KE, Straus SE, Wang H, Wright PF, Pachucki CT, Gershon AA, Arbeit RD, Davis LE, Simberkoff MS, Weinberg A, Williams HM, Cheney C, Petrukhin L, Abraham KG, Shaw A, Manoff S, Antonello JM, Green T, Wang Y, Tan C, Keller PM; Shingles Prevention Study Group. A real-time PCR assay to identify and discriminate among wild-type and vaccine strains of varicella-zoster virus and herpes simplex virus in clinical specimens, and comparison with the clinical diagnoses. J Med Virol. 2009 Jul;81(7):1310-22. doi: 10.1002/jmv.21506. PMID 19475609
- [Result] Weinberg A, Zhang JH, Oxman MN, Johnson GR, Hayward AR, Caulfield MJ, Irwin MR, Clair J, Smith JG, Stanley H, Marchese RD, Harbecke R, Williams HM, Chan IS, Arbeit RD, Gershon AA, Schodel F, Morrison VA, Kauffman CA, Straus SE, Schmader KE, Davis LE, Levin MJ; US Department of Veterans Affairs (VA) Cooperative Studies Program Shingles Prevention Study Investigators. Varicella-zoster virus-specific immune responses to herpes zoster in elderly participants in a trial of a clinically effective zoster vaccine. J Infect Dis. 2009 Oct 1;200(7):1068-77. doi: 10.1086/605611. PMID 19712037
- [Result] Schmader KE, Oxman MN, Levin MJ, Johnson G, Zhang JH, Betts R, Morrison VA, Gelb L, Guatelli JC, Harbecke R, Pachucki C, Keay S, Menzies B, Griffin MR, Kauffman C, Marques A, Toney J, Keller PM, Li X, Chan IS, Annunziato P; Shingles Prevention Study Group. Persistence of the efficacy of zoster vaccine in the shingles prevention study and the short-term persistence substudy. Clin Infect Dis. 2012 Nov 15;55(10):1320-8. doi: 10.1093/cid/cis638. Epub 2012 Jul 24. PMID 22828595
- [Result] Schmader KE, Johnson GR, Saddier P, Ciarleglio M, Wang WW, Zhang JH, Chan IS, Yeh SS, Levin MJ, Harbecke RM, Oxman MN; Shingles Prevention Study Group. Effect of a zoster vaccine on herpes zoster-related interference with functional status and health-related quality-of-life measures in older adults. J Am Geriatr Soc. 2010 Sep;58(9):1634-41. doi: 10.1111/j.1532-5415.2010.03021.x. PMID 20863322
- [Result] Morrison VA, Oxman MN, Levin MJ, Schmader KE, Guatelli JC, Betts RF, Gelb LD, Pachucki CT, Keay SK, Menzies B, Griffin MR, Kauffman CA, Marques AR, Toney JF, Simberkoff MS, Serrao R, Arbeit RD, Gnann JW, Greenberg RN, Holodniy M, Keitel WA, Yeh SS, Davis LE, Crawford GE, Neuzil KM, Johnson GR, Zhang JH, Harbecke R, Chan IS, Keller PM, Williams HM, Boardman KD, Silber JL, Annunziato PW; Shingles Prevention Study Group. Safety of zoster vaccine in elderly adults following documented herpes zoster. J Infect Dis. 2013 Aug 15;208(4):559-63. doi: 10.1093/infdis/jit182. Epub 2013 Apr 30. PMID 23633406
- See also: Related Info — http://www.research.va.gov/programs/csrd/csp.cfm